CLINICAL TRIAL: NCT04477109
Title: Effectiveness of Low Level Laser Therapy on Insulin Resistance and Inflammatory Biomarkers in Obese Postmenopausal Breast Cancer Risk Women
Brief Title: Effectiveness of Low Level Laser Therapy on Insulin Resistance and Inflammatory Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P.T.REC/012/002677
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Insulin Resistance; Inflammatory Markers
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level laser in addition to diet recommendations (Active Comparator): The laser consists of a semiconductor and operates at a wavelength of 650 nanometre. The laser installed in the watch comprises 10 individual laser beams for the wrist and an additional adapter for nasal stimulation. The output power is 5 megawatt, but it can also be adjusted. The device operates at an ambient temperature of -20 to +40 ° C and a relative humidity of ≤ 85%. The laser watch can be used for a variable irradiation period of 10-60 min. the device will be applied on specific acupuncture points (N acupuncture point, Radial artery acupuncture points, and ulnar artery acupuncture points) combined with nasal laser irradiation at the same time, once per day, 3 times per week for three months
  Interventions: Device: low level laser in addition to diet recommendations
- sham laser application in addition to diet recommendations (Sham Comparator): while the control group will stick to the same line of treatment but with sham laser application
  Interventions: Other: sham laser application in addition to diet recommendations

INTERVENTIONS:
Device: low level laser in addition to diet recommendations — The laser consists of a semiconductor and operates at a wavelength of 650 nanometre. The laser installed in the watch comprises 10 individual laser beams for the wrist and an additional adapter for nasal stimulation. The output power is 5 megawatt
  Arms: low level laser in addition to diet recommendations
Other: sham laser application in addition to diet recommendations — sham laser application in addition to diet recommendations
  Arms: sham laser application in addition to diet recommendations

SUMMARY:
It is an interventional study in which 60 women estimated to enroll according to random allocation and assigned into two groups equal. The study group will receive active low level laser in addition to diet recommendations while the control group will stick to the same line of treatment but with sham laser application. The laser consists of semiconductor and operates at a wavelength of 650 nanometre. The laser installed in the watch comprises 10 individual laser beams for the wrist and an additional adapter for nasal stimulation. The output power is 5 megawatt, but it can also be adjusted. The device operates at an ambient temperature of -20 to +40 ° C and a relative humidity of ≤ 85%. The laser watch can be used for a variable irradiation period of 10-60 min. the device will be applied on specific acupuncture points (N acupuncture point, Radial artery acupuncture points, and ulnar artery acupuncture points) combined with nasal laser irradiation at the same time, once per day, 3 times per week for three months

DETAILED DESCRIPTION:
PURPOSE:

To determine the effectiveness of low level laser therapy on insulin resistance and inflammatory biomarkers in obese postmenopausal breast cancer risk women

BACKGROUND:

The American Obesity Association (2002, 2003) defines obesity as 'a complex, multifactorial chronic disease involving environmental (social and cultural), genetic, physiologic, metabolic, behavioral, and psychological components'. However, the most commonly used definitions of obesity are based on BMI, which is defined as weight in kilograms divided by height in meters squared. In adults, obesity is generally defined as a BMI of 30.0 or greater. Obesity has become a major contributor to the global burden of chronic disease and disability. It is a complex condition with serious social and psychological dimensions, affecting virtually all ages and socioeconomic group Obesity is associated with an increased risk of developing insulin resistance and type 2 diabetes. In obese individuals, adipose tissue releases increased amounts of non-esterified fatty acids, glycerol, hormones, proinflammatory cytokines and other factors that are involved in the development of insulin resistance. In overweight and obesity, there exists low-grade chronic inflammation characterized by the increase of cytokines and serum concentrations such as fibrinogen and C-reactive protein (CRP) The areas of low - intensity laser use have expanded in several conditions by different mechanisms and ways. LLLT has been used as an important tool for the control of the inflammatory process. Its anti-inflammatory effect has been studied and its ability to induce analgesia under different conditions has also been reported. Because laser acupuncture appears to be safe, it could be considered as a complementary form of palliative care for prevention of cancer risk, especially for clinical problems for which conventional care options are limited. Investigations suggest the benefits of low-level laser therapy (LLLT) to improve noninvasive body contouring treatments, inflammation, insulin resistance and to reduce body fat.

HYPOTHESES:

Low level laser therapy in form of laser watch has no effect on insulin resistance inflammatory biomarkers in obese postmenopausal breast cancer risk women

RESEARCH QUESTION:

Does low level laser therapy has an effect on insulin resistance inflammatory biomarkers in obese postmenopausal breast cancer risk women?

ELIGIBILITY:
Inclusion Criteria:

* • Sixty Postmenopausal women (60-75 y)

  * Body mass index (BMI) ranged from 30 to 34.9 kg/m2
  * Family history of breast cancer

Exclusion Criteria:

* • women receiving weight-reduction interventions

  * taking lipid lowering drugs
  * regular medications(e.g., β-blockers, α-blockers, digoxin, diuretics, aspirin, nitrates, or hormones)
  * having active chronic illness (e.g., rheumatoid arthritis, hyperthyroidism, and inflammatory bowel disease)
  * cognitive impairment that will make it difficult to partake in the study
  * presence of malignant disease
  * blood donation within the last 30 days
  * Participation as a subject in any type of study or research during the prior 90 days

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 12 weeks
  change of insulin resistance by Homeostatic Model Assessment of Insulin Resistance
inflammatory markers | 12 weeks
  change of inflammatory markers(C-reactive protein-erythrocyte sedimentation rate-White blood cells-lymphocytes)

SECONDARY OUTCOMES:
body mass index | 12 weeks
  divide weight by height square

CONTACTS AND LOCATIONS:
Overall Officials: marwa m elsayed, phd, Principal Investigator — lecturer at physical therapy faculty cairo university
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: one year after completing the study
Access Criteria: journal publishing the study
URL: http://Scholar.cu.edu.eg/p_t